CLINICAL TRIAL: NCT07288749
Title: Efficacy Evaluation of Glimepiride in Patients With Type 2 Diabetes Mellitus and Chronic Heart Failure With Reduced Ejection Fraction: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial.
Brief Title: Efficacy Evaluation of Glimepiride in Patients With Type 2 Diabetes Mellitus and Chronic Heart Failure With Reduced Ejection Fraction.
Acronym: GLID-HF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Nanjing Medical University (Other); Second Xiangya Hospital of Central South University (Other); Huaxi Hospital (Other); Zhongnan Hospital (Other); Xiangya Hospital (Other); Beijing Anzhen Hospital (Other); The First Affiliated Hospital of Air Force Medicial University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Anhui Provincial Hospital (Other Government); Southwest Medical University (Other); First Hospital of China Medical University (Other); Wuhan Central Hospital (Other); Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Prof., Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJ-GLID-HF
Record Dates: First submitted 2025-12-05; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Chronic Heart Failure (CHF)
Keywords: Type 2 Diabetes Mellitus (T2DM); Chronic heart failure (CHF); Glimepiride; Randomized clinical trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employed a double-blind design, meaning that neither the patients, investigators, study coordinators, members of the endpoint adjudication committee, nor the data analysts were aware of the specific group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glimepiride group (Experimental): Standardized treatment for chronic heart failure + standardized treatment for type 2 diabetes + oral glimepiride (initial oral dose is 2 mg once daily. After 4 weeks, adjust the oral dose based on glycemic control and tolerability: If glycemic control is adequate, maintain the initial oral dose. If glycemic control is inadequate, modify the oral dose to 4 mg once daily.)
  Interventions: Drug: Glimepiride (oral)
- Placebo group (Placebo Comparator): Standardized treatment for chronic heart failure + standardized treatment for type 2 diabetes + oral placebo (equivalent placebo administered according to the same regimen)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glimepiride (oral) — Standardized treatment for chronic heart failure + standardized treatment for type 2 diabetes + oral glimepiride (initial oral dose is 2 mg once daily. After 4 weeks, adjust the oral dose based on glycemic control and tolerability: If glycemic control is adequate, maintain the initial oral dose. If glycemic control is inadequate, modify the oral dose to 4 mg once daily.)
  Arms: Glimepiride group
Drug: Placebo — Standardized treatment for chronic heart failure + standardized treatment for type 2 diabetes + oral placebo (equivalent placebo administered according to the same regimen)
  Arms: Placebo group

SUMMARY:
Evaluating the safety and efficacy of glimepiride in patients with type 2 diabetes and chronic heart failure with reduced ejection fraction--a multicenter randomized controlled study.

DETAILED DESCRIPTION:
Diabetes and heart failure share common pathophysiological mechanisms. The synergistic effects of managing both conditions, along with the potential for diabetes treatment to modulate the risk of heart failure outcomes, hold significant medical promise.Currently, the relationship between sulfonylureas，primarily including glimepiride, and heart failure outcomes remains poorly understood, with ongoing controversy regarding their cardiovascular effects in observational studies. No large-scale, randomized controlled trials have yet been conducted to validate the impact of sulfonylureas on patients with established heart failure. Our prospective cohort studies have preliminarily confirmed the cardioprotective effects of glimepiride in patients with type 2 diabetes complicated by chronic heart failure, demonstrating a favorable safety profile. Therefore, this study aims to conduct a prospective, multicenter, randomized, double-blind, placebo-controlled clinical trial to evaluate the therapeutic efficacy of glimepiride in patients with type 2 diabetes complicated by chronic heart failure.This study plan aims to recruit 1,484 eligible participants, who will be randomly assigned in a 1:1 ratio to either the glimepiride group or the placebo group. The total study duration is 36 months, with all participants required to complete baseline visits and outpatient follow-ups at months 1, 3, 6, 9, 12, 18, 24, 30 and 36.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old at the time of enrollment; gender is not restricted.
2. Patients diagnosed with type 2 diabetes according to the "Chinese Diabetes Prevention and Management Guidelines (2024 Edition)" issued by the Chinese Medical Association Diabetes Branch, with a confirmed diagnosis at least three months prior.
3. According to the "Chinese Guidelines for the Diagnosis and Treatment of Heart Failure (2024 Edition)" issued by the Chinese Society of Cardiology, the diagnosis is heart failure with reduced ejection fraction (HFrEF) or heart failure with mildly reduced ejection fraction (HFmrEF), confirmed at least three months prior.
4. NYHA heart failure classification stage II-IV;
5. Within 12 months prior to enrollment, left ventricular ejection fraction (LVEF) was < 50%, as determined by echocardiography, nuclear ventriculography, angiography, or cardiac magnetic resonance imaging.
6. NT-proBNP levels ≥ 600 pg/mL in patients with no recent hospitalization for heart failure; NT-proBNP levels ≥ 400 pg/mL within the past 12 months due to heart failure hospitalization; NT-proBNP levels ≥ 900 pg/mL in patients with heart failure complicated by atrial fibrillation/flutter.
7. Patients must have experienced stable heart failure symptoms for at least three months prior to enrollment and must have received standardized chronic heart failure therapy and guideline-directed diabetes management for no less than two weeks before enrollment, with no dose adjustments during this period.
8. Participation is voluntary and requires signing an informed consent form; follow-up can extend beyond three years.

Exclusion Criteria:

1. Heart failure caused by valvular disease, congenital heart conditions, pericardial diseases, arrhythmias, or non-cardiogenic illnesses; as well as heart failure resulting from failure of vital organs such as renal or hepatic failure; and right-sided heart failure due to pulmonary origin or other definitive causes.
2. Currently experiencing acute decompensated heart failure (ADHF) or hospitalized for ADHF within the previous four weeks before enrollment.
3. Patients scheduled to undergo coronary artery revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass grafting [CABG]) or cardiac resynchronization therapy following randomization, or who have received cardiac resynchronization therapy within 12 weeks prior to enrollment.
4. Any conditions other than cardiovascular diseases, including but not limited to malignancies with an expected survival of less than three years, severe mental disorders, hematologic diseases, neuroendocrine disorders, elevated liver transaminases and alkaline phosphatase levels exceeding three times the upper limit of normal (ULN), renal impairment indicated by serum creatinine greater than 2 mg/dL (176.82 µmol/L), and hyperkalemia with serum potassium levels exceeding 5.5 mmol/L.
5. Chronic kidney disease stage 3b or more advanced renal impairment (i.e., estimated glomerular filtration rate [eGFR]/creatinine clearance [CrCl] <45 ml/min);
6. Left ventricular outflow tract obstruction, acute or fulminant myocarditis, aortic aneurysm, aortic dissection, or significant hemodynamic changes caused by unrepaired valves;
7. Cardiac shock, uncontrollable malignant arrhythmias, second-degree or higher sinus or atrioventricular block without pacemaker therapy, progressive unstable angina pectoris, or acute myocardial infarction;
8. Uncontrolled hypertension with systolic blood pressure (SBP) ≥180 mmHg and/or diastolic blood pressure (DBP) ≥110 mmHg; or SBP <90 mmHg and/or DBP <60 mmHg;
9. Female patients who are pregnant, planning to become pregnant, or breastfeeding;
10. Patients who have participated in any other investigational medicinal product clinical trial within the past 4 weeks;
11. Patients with a history of allergies or hypersensitivity to glimepiride or its derivatives;
12. Received glimepiride treatment within 8 weeks prior to enrollment or previously demonstrated intolerance to glimepiride;
13. Patients refusing to comply with study requirements to complete the research;
14. Conditions where the investigator deems the patient unable to understand and/or comply with study medications, procedures, or any other circumstances that may prevent completion of the study;
15. Any other reason deemed inappropriate for inclusion by the study physician.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1484 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite endpoint of cardiovascular death, heart transplantation, or worsening heart failure (defined as rehospitalization for heart failure or an emergency heart failure visit requiring intravenous therapy). | 3 years
  The Primary Outcome is defined as a composite endpoint consisting of the time to the first occurrence of any of the following events:
  1. Cardiovascular death is defined as any death due to a direct cardiovascular cause.
  2. Heart transplantation is defined as receiving an allogeneic in situ heart transplant due to end-stage heart failure. The event date is defined as the date of surgery.
  3. Heart failure exacerbation is defined as requiring intensive treatment due to worsening symptoms and signs of heart failure, meeting any of the following criteria: ① readmission for heart failure; ② urgent heart failure visit requiring intravenous therapy.

SECONDARY OUTCOMES:
All-cause mortality rate | 3 years
  Death occurring during the study period for any cause. This is the most objective and unbiased endpoint. All deaths, whether cardiovascular-related or not, are included in this endpoint.
Cardiovascular death, heart transplantation, or readmission due to heart failure | 3 years
  Time to the first occurrence of any of the following events: cardiovascular death, heart transplantation, or rehospitalization for heart failure (defined as the primary endpoint).
Cardiovascular death, heart transplantation | 3 years
  Time to the first occurrence of any of the following events: cardiovascular death or heart transplantation (defined as the primary endpoint).
Rehospitalization due to heart failure | 3 years
  Time to first rehospitalization due to heart failure (defined as the primary endpoint).
Incidence of discontinuing treatment due to worsening heart failure | 3 years
  The patient or their family voluntarily decides to forgo aggressive life-sustaining treatment-including intravenous medications, mechanical ventilation, and renal replacement therapy-due to the extremely poor prognosis of heart failure, inability to tolerate treatment, or other reasons, ultimately resulting in the patient's death after treatment is discontinued.
Rate of successful resuscitation following cardiac arrest | 3 years
  An event where spontaneous circulation is successfully restored for ≥20 minutes following cardiac arrest (defined as pulseless ventricular tachycardia, ventricular fibrillation, or pulseless electrical activity) through cardiopulmonary resuscitation (including defibrillation, external chest compressions, pharmacotherapy, etc.).
Incidence of malignant arrhythmias | 3 years
  Clinically significant ventricular arrhythmias confirmed by electrocardiogram, Holter monitoring, or implantable device recordings. Typically includes: sustained ventricular tachycardia (lasting ≥30 seconds or requiring urgent termination due to hemodynamic instability); ventricular fibrillation; ventricular arrhythmias resulting in appropriate electrical therapy (applicable to patients with implantable cardioverter-defibrillators [ICDs] or cardiac resynchronization therapy defibrillators [CRT-Ds]).
Rate of serum NT-proBNP decrease | 3 years
  The relative rate of change in serum NT-proBNP levels from baseline to a predetermined study time point (e.g., 3 months, 6 months, or 12 months). Calculation formula: (Follow-up value - Baseline value) / Baseline value × 100%.
Changes in Kansas Cardiomyopathy Questionnaire (KCCQ) scores | 3 years
  The absolute change in the KCCQ overall summary score (or domain-specific scores such as physical function, symptom frequency, quality of life, and social limitations) from baseline to a predetermined study time point (e.g., 3 months, 6 months, or 12 months). Calculation Method: Follow-up score - Baseline score.
Changes in 6-Minute Walk Test (6MWT) Results | 3 years
  Change in 6-minute walk distance (6MWD) from baseline to follow-up (in meters).
Incidence of non-fatal myocardial infarction or non-fatal stroke | 3 years
  Time to the first occurrence of either a non-fatal myocardial infarction or a non-fatal stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hostipal, Wuhan, Hubei, China

REFERENCES:
- [Result] Karwi QG, Ho KL, Pherwani S, Ketema EB, Sun Q, Lopaschuk GD. Corrigendum to: Concurrent diabetes and heart failure: interplay and novel therapeutic approaches. Cardiovasc Res. 2022 Jun 22;118(7):1850. doi: 10.1093/cvr/cvab355. No abstract available. PMID 34897419
- [Result] Fitchett DH, Udell JA, Inzucchi SE. Heart failure outcomes in clinical trials of glucose-lowering agents in patients with diabetes. Eur J Heart Fail. 2017 Jan;19(1):43-53. doi: 10.1002/ejhf.633. Epub 2016 Sep 21. PMID 27653447
- [Result] He W, Yuan G, Han Y, Yan Y, Li G, Zhao C, Shen J, Jiang X, Chen C, Ni L, Wang DW. Glimepiride Use is Associated with Reduced Cardiovascular Mortality in Patients with Type 2 Diabetes and Chronic Heart Failure: A Prospective Cohort Study. Eur J Prev Cardiol. 2022 Dec 27:zwac312. doi: 10.1093/eurjpc/zwac312. Online ahead of print. PMID 36573717